CLINICAL TRIAL: NCT00164476
Title: Promoting Prevention Among Adults With Disabilities
Brief Title: Promoting Clinical Preventive Services Among Adults With Disabilities
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCBDDD-CCR323280
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2005-09-14 (Estimated); Status verified 2005-09

CONDITIONS: Physical Disability
MeSH Terms: interventions — Control Groups

INTERVENTIONS:
Behavioral: Preventive Services Prevention Kit
Behavioral: peer mentors (control group)

SUMMARY:
Project SHIELD (Strategies and health Interventions to Enhance Life with Disability) is a participatory action research project to test an intervention package combining a resource kit with peer mentoring in improving consumer education about primary preventive services

DETAILED DESCRIPTION:
Adults with disabilities use primary preventive health care services (basic screenings, immunizations, and hevior health counseling) at rates below those recommended by the US Preventive Services Task Force and Healthy People 2010. This projects is to carry out a community-based campaign to increase preventive care knowledge and service use among adults with physical disabilities. Focus group methodology will be used to determine the specific preventive service priorities of the disability community so that targeted resource materials for consumers and physicians can be developed. Second, a randomized control group experiment will be implemented to evaluate the effectiveness of the targeted resource materials, followed by dissemination of the Preventive Services Resource Kits.

ELIGIBILITY:
Inclusion Criteria:

* primary residence in Northern Virginia presence of a physical disability at least 18 years old

Exclusion Criteria:

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2003-10; Study Completion 2005-06

PRIMARY OUTCOMES:
Prevention-related knowledge and beliefs
Self-efficacy
Service-seeking intent
Service utilization

SECONDARY OUTCOMES:
perceptions of the Preventive Service Resource Kit

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne L Groah, MD, Principal Investigator — Medstar Health Research Institute
Locations (1):
- National Rehabilitation Hospital, Washington D.C., District of Columbia, United States